CLINICAL TRIAL: NCT00422981
Title: A Phase 2, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Effect on Cognitive Function of AL-108 After 12 Weeks of Intranasal Administration in Subjects With Mild Cognitive Impairment
Brief Title: Safety, Tolerability and Efficacy Study to Evaluate Subjects With Mild Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL-108-211
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Mild Cognitive Impairment, So Stated
Keywords: Dementia; Memory; Alzheimers; Cognition; Mind; Aging
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — davunetide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AL-108 5 mg (Active Comparator): 5 mg QD
  Interventions: Drug: AL-108
- AL-108 15 mg (Active Comparator): 15 mg BID
  Interventions: Drug: AL-108
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AL-108 — 5 mg QD
  Arms: AL-108 5 mg
Drug: AL-108 — 15 mg BID
  Arms: AL-108 15 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if different doses of Investigational Drug are safe, tolerable, and if they have an effect on Mild Cognitive Impairment (MCI).

DETAILED DESCRIPTION:
Pre-Clinical experiments indicate the AL-108 compound has neuroprotective, cognitive protective and neurotrophic properties; therefore, the compound could be tested in a variety of human diseases. Human diseases include Cognitive impairment associated with aging or neurodegenerative diseases such as Alzheimer's Disease.

This clinical trial aims at providing the dose rationale as well as safety and tolerability information for AL-108 as evaluated after 12 weeks of intranasal administration in subjects with Mild Cognitive Impairment (MCI).

There are currently no drugs approved for the treatment of MCI nor accepted treatment or standard treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female, at 55-85 years of age (inclusive) at screening
* Self-reported memory complaint, corroborated by spouse or companion as appropriate.
* Wechsler Memory Scale III (WMS-III) age-adjusted Logical Memory II score ≤ 5.
* Mini-Mental State Exam (MMSE) ≥24.
* Center for Epidemiologic Studies-Depression (CES-D) score <27.
* Normal thyroid function, defined as TSH, T3 and T4 within normal limits.
* Agree not to consume alcoholic beverages within 8 hours of each study visit.
* Willing and able to sign informed consent and complete the CTB and all other tests and procedures as listed in the protocol.
* Fluently reads and speaks English.
* Female subjects must be surgically sterile or post-menopausal for at least 2 years. If <2 years post-menopausal, then a follicle stimulating hormone (FSH) ≥40 mIU/mL must be obtained.

Exclusion Criteria:

* Subjects who have any significant, untreated psychiatric illness or any CNS condition (such as schizophrenia, Parkinson's disease, stroke, etc.) that could interfere with the study evaluations or procedures or which poses an additional risk. Subjects with a history of uncomplicated depression may participate if in remission and on a stable dose of antidepressant medication for at least 2 months.
* History of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.
* History of alcohol or substance abuse or dependence within the past year.
* Acute infective sinusitis.
* History or presence of an abnormality of the external or internal structures of the nose or nasopharynx, except for surgical correction of the nasal septum or a "broken nose" at least 2 years previously, or surgical repair of cleft palate when <30 years of age.
* Use of medications that are known to cause frank obtundation of cognition
* Use of any approved or investigational medication for Alzheimer's Disease within 3 months of screening
* History of or current significant systemic disease judged to interfere with the study evaluations or likely to be a safety concern.
* Untreated sleep apnea or treatment for sleep apnea for <3 months.
* Abnormal clinical laboratory test results, specifically: Alanine transaminase (ALT) or aspartate transaminase (AST) >2 х the upper limit of normal (ULN),Hematology <80% the lower limit of normal, Creatinine ≥2 mg/dL and ,Other clinical laboratory values or vital signs considered clinically significant in the opinion of the Investigator.
* Treatment with any investigational drug, biologic, or device within the previous 30 days prior to screening.
* Surgery involving general anesthesia within the past 3 months or planned surgery requiring general anesthesia during the study period.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 12 on the Composite Memory Variable | 12 weeks

SECONDARY OUTCOMES:
Changes in the Composite Memory Variable from baseline to weeks 4, 8, and 16 | 16 weeks
Changes in test battery individual items from baseline to endpoints (weeks 4, 8, 12, and 16). | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donald E Schmechel, MD, Principal Investigator — Memory Assessment and Research Services
Locations (17):
- United States (17):
  - Pivotal Research, Peoria, Arizona
  - Collaborative Neuroscience Network, Garden Grove, California
  - Synergy Research, National City, California
  - Pacific Research Network, Inc, San Diego, California
  - Meridien Research, Brooksville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Meridien Research, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Clinical Research Center of Indian River Medical Center, Vero Beach, Florida
  - Comprehensive Neuroscience, Hoffman Estates, Illinois
  - The Memory Enhancement Center of America, Long Branch, New Jersey
  - SPRI Clinical trials, Brooklyn, New York
  - Memory Assessment and Research Services, Wilmington, North Carolina
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Senior Adults Speciality Research, Austin, Texas

REFERENCES:
- [Derived] Gozes I, Blatt J, Lobyntseva A. Davunetide sex-dependently boosts memory in prodromal Alzheimer's disease. Transl Psychiatry. 2024 Oct 2;14(1):412. doi: 10.1038/s41398-024-03118-0. PMID 39358355
- [Derived] Morimoto BH, Schmechel D, Hirman J, Blackwell A, Keith J, Gold M; AL-108-211 Study. A double-blind, placebo-controlled, ascending-dose, randomized study to evaluate the safety, tolerability and effects on cognition of AL-108 after 12 weeks of intranasal administration in subjects with mild cognitive impairment. Dement Geriatr Cogn Disord. 2013;35(5-6):325-36. doi: 10.1159/000348347. Epub 2013 Apr 13. PMID 23594991